CLINICAL TRIAL: NCT00395278
Title: Development of Serologic Assays for Human Herpes Virus-8
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 999907018; 07-CC-N018
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Kaposi Sarcoma; HIV Infection
Keywords: Antibody; Kaposi's Sarcoma; HIV; Kaposi Sarcoma
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- HIV negative: HIV negative without Kaposi sarcoma
- HIV positive: HIV positive without Kaposi sarcoma
- HIV positive KS: HIV positive with Kaposi sarcoma

SUMMARY:
Dr. Burbelo and colleagues have developed a technique for rapidly and quantitatively detecting antibody responses in sera to a variety of pathogens using recombinant proteins. We would like to apply this technique to develop an assay for detecting antibodies to HHV-8 (KSHV, the etiologic agents of Kaposi's sarcoma, an AIDS-defining condition). We initially plan to examine samples from patients with Kaposi's sarcoma, since all those patients are almost certainly infected with HHV-8. We are thus using samples from patients with previously diagnosed Kaposi's sarcoma. The samples in question are stored at the NCI FCRF repository operated by SAIC Frederick or in Rockville, MD.

DETAILED DESCRIPTION:
Our colleagues have developed a technique for rapidly and quantitatively detecting antibody responses in sera to a variety of antigens using recombinant proteins. We would like to apply this technique to develop an assay for detecting antibodies to HHV- 8 (KSHV, the etiologic agent of Kaposi s sarcoma, an AIDS-defining condition). In addition we would like to potentially measure antibody responses to HIV, other infectious agents, and human antigens, to see if antibodies (or high antibody titers) to these antigens are associated with Kaposi s sarcoma or HIV infection. We initially plan to examine samples from patients with Kaposi s sarcoma, since all those patients are almost certainly infected with HHV-8. We would subsequently plan to examine samples from HIV positive and HIV negative patients without known Kaposi s sarcoma. We are thus requesting permission to use samples from patients with and without previously diagnosed Kaposi's Sarcoma. In addition to antibody testing, we would also like to examine these samples for evidence of infection with other infectious agents, such as newly identified or unknown viruses, using techniques such as PCR or deep

sequencing.

ELIGIBILITY:
* Data analysis only

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stored samples from individuals who had previously participated in studies conducted by the NIAID CCMD HIV/AIDS program
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2006-10-30 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
HHV8 serology | At sample collection
  Direction of antibodies to HHV8 proteins

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Kovacs, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States